CLINICAL TRIAL: NCT01086111
Title: Mechanisms of Type 2 Diabetes Improvement, Besides Weightloss After Gastric Bypass
Brief Title: The Effect of a Gastric Bypass on Type 2 Diabetes in the Morbidly Obese Patient
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Matthias Lannoo, medical doctor, University Hospital, Gasthuisberg
Other Study IDs: S51169
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Type 2 Diabetes; Morbid Obesity
Keywords: type 2 diabetes; gastric bypass; sleeve gastrectomy; clamp study; weight loss surgery
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- PMSF: type 2 diabetes patient receiving a protein sparing diet
- sleeve gastrectomy: type 2 diabetes patient receiving a gastric bypass
- RYGBP: type 2 diabetes patient receiving a gastric bypass

SUMMARY:
Proof of concept, of RYGBP and its capabilities to cure type 2 diabetes (DM 2) and sleep apnea has already been recognized in the reports on weight loss surgery.

The investigators project aims to prove that RYGBP also recovers the beta cell function (BCF) Clamp tests, the gold standard for testing IS and BCF, will be performed preoperative and early postoperatively.

Aims & methodology:

Analysis of the short-term effect of gastric bypass and sleeve gastrectomy on insulin sensitivity and beta cell function.

Preoperative baseline insulin sensitivity and beta cell function will be assessed with euglycemic and hyperglycemic clamp tests. These results will be compared with the results of the same tests carried out 3 weeks postoperative.

To determine if the duodenal exclusion is causing this effect. The results of the clamp tests 3 weeks postoperative will be compared

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 18 to 65
* BMI > 35 kg/m2
* Subject is capable and willing to give informed consent.
* In the surgical groups indication for surgery is approved by the local multidisciplinary obesity workgroup following the NIH guidelines of 199112.
* Patient suffers from type 2 diabetes necessitating insulin therapy.
* Subject is a non-smoker for at least 6 months prior to study start.
* Female patients of child bearing potential must use oral, injected or implanted hormonal methods of contraception from at least the commencement of their last normal period prior to the screening visit. Patients using hormonal contraception should use a barrier method in addition from screening visit until their next normal period following the end of the study.
* Female patients of non-child bearing potential defined as:

  * Post-menopausal females, being amenorrhoeic for at least 1 year
  * Pre-menopausal females with a documented hysterectomy or bilateral oophorectomy.

Exclusion Criteria:

* Female patient is pregnant or breastfeeding.
* BMI < 35 kg/m2
* Patient suffers from an endocrine disease, besides diabetes and thyroid disease, such as Cushing's disease, Addison's disease, hypothalamic tumor…)
* Patient suffers from type 1 diabetes, MODY or LADA
* Patient has undergone previous surgical procedure for weight loss
* Patient is considered ASA 4 or more according to the ASA physical status classification system of the American Society of Anesthesiologists.
* Patient suffers from liver cirrhosis
* Patient uses steroids
* Patient uses cyclosporin
* Recent (<30 days) or simultaneous participation in another clinical trial.
* Any situation that can compromise the study, including serious illness or a predictable lack of cooperation from the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type 2 diabetes patients with a BMI > 35kg/m²
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity and beta cell function | 3 weeks
  insulin sensitivity and beta cell function changes 3 weeks after RYGB, sleeve gastrectomy and protein sparing diet using euglycaemic and hyperglycemic clamp techniques.

SECONDARY OUTCOMES:
changes in plasma levels of gut hormones and inflammation markers | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, gasthuisberg, Leuven, Belgium